CLINICAL TRIAL: NCT05456555
Title: The Flapless Approach With and Without Enamel Matrix Derivatives in the Regenerative Treatment of Intrabony Defects: a Randomized Controlled Clinical Trial
Brief Title: The Flapless Approach in Periodontal Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMDTurin1
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis, Adult; Intrabony Periodontal Defect
MeSH Terms: conditions — Chronic Periodontitis | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flapless with Enamel Matrix Derivatives (EMD) (Experimental): Closed non-surgical treatment of periodontal intrabony defects with the combined use of Enamel Matrix Derivatives (EMD).
  Interventions: Procedure: Flapless with Enamel Matrix Derivatives (EMD)
- Flapless alone (Active Comparator): Closed non-surgical treatment of periodontal intrabony defects without any adjunct.
  Interventions: Procedure: Flapless without Enamel Matrix Derivatives (EMD)

INTERVENTIONS:
Procedure: Flapless with Enamel Matrix Derivatives (EMD) — Experimental sites will receive a closed non-surgical treatment with a combined use of minicurettes and ultrasonic instruments with thin and delicate tips. Teeth will be instrumented until no residual calculus could be detected. A visualization of the root surface will be accomplished under magnification by using dental loups 4.0X. In the test group, the roots will be conditioned with 24% ethylenediaminetetraacetic acid (EDTA) for 2 minutes. After rinsing with sterile saline, enamel matrix derivatives (EMD) will be applied on the dried root surface.
  Arms: Flapless with Enamel Matrix Derivatives (EMD)
Procedure: Flapless without Enamel Matrix Derivatives (EMD) — Experimental sites will receive a closed non-surgical treatment with a combined use of minicurettes and ultrasonic instruments with thin and delicate tips. Teeth will be instrumented until no residual calculus could be detected. A visualization of the root surface will be accomplished under magnification by using dental loups 4.0X. No adjunct will be administered.
  Arms: Flapless alone

SUMMARY:
The present investigation is designed in order to compare the radiographic and clinical effectiveness of flapless procedure performed alone or in combination with enamel matrix derivatives in the periodontal regenerative treatment of deep intrabony defects in patients with moderate or severe periodontitis. The study will have a follow-up of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of periodontitis stage III or IV;
* presence of at least one tooth with ≥6 mm associated with a radiographic intrabony defect ≥3 mm at least 2 months after the completion of non-surgical therapy;
* a full-mouth plaque score and full-mouth bleeding score <15% at the time of the experimental procedure;
* signed informed consent.

Exclusion Criteria:

* relevant medical disorders contraindicating periodontal surgery or detrimental to periodontal healing;
* consumption of drugs known to affect periodontal status;
* pregnancy and lactation;
* third molars, teeth with furcation involvement or inadequate endodontic treatment and/or prosthetic restoration;
* heavy smokers >10 cigarettes per day.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change | 12 months
  Clinical attachment level will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

SECONDARY OUTCOMES:
Radiographic bone level change | 12 months
  Periapical standardized radiographs will be taken by a clinician masked to the clinical measurements using the paralleling technique and individually customized bite-blocks (RINN XCP Film Holding Instruments, Dentsply, York, USA)
Probing pocket depth change | 12 months
  Probing depth will be assessed on the experimental teeth using periodontal probe (PCP 15/11.5, Hu-Friedy, Chicago, IL, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aimetti M, Stasikelyte M, Mariani GM, Cricenti L, Baima G, Romano F. The flapless approach with and without enamel matrix derivatives for the treatment of intrabony defects: A randomized controlled clinical trial. J Clin Periodontol. 2024 Sep;51(9):1112-1121. doi: 10.1111/jcpe.14028. Epub 2024 Jun 10. PMID 38859627